CLINICAL TRIAL: NCT06260072
Title: Magnesium and Riboflavin Treatment for Post-Concussion Headache
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Stephanie Hartman, MD, Associate Director of Primary Care UVA Student Health & Wellness, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-HSR 21920
Record Dates: First submitted 2024-02-06; First posted 2024-02-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Concussion, Intermediate
Keywords: Concussion; Headache
MeSH Terms: conditions — Brain Concussion; Headache | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active study product (Active Comparator): 400 mg of Magnesium Oxide and 400 mg Riboflavin in capsule formation
  Interventions: Drug: magnesium and riboflavin supplement
- Placebo study product (Placebo Comparator): Inert placebo in capsule formation
  Interventions: Drug: magnesium and riboflavin supplement

INTERVENTIONS:
Drug: magnesium and riboflavin supplement — Five capsules considered one dose of the intervention (one 400 mg magnesium capsule and four 100 mg riboflavin capsules)

SUMMARY:
This clinical trial will try to determine if the supplements magnesium and riboflavin will reduce the pain and duration of headaches in persons diagnosed with a concussion. The participant will be randomized to either active magnesium and riboflavin capsules or placebo (inert) capsules. The capsules will be taken once a day for 14 days. The participant will also complete a short diary form for the 14 days and will have 3 follow up visits either by telephone or in person.

ELIGIBILITY:
Inclusion Criteria:

* Seen at University of Virginia Student Health and Wellness Center or Emergency Department for Initial Visit for Concussion;
* Less than 3 days have elapsed since their injury;
* Able to swallow capsules

Exclusion Criteria:

* Concussion complicated by cranial bleed, skull fracture, additional severe injury;
* Kidney disfunction or failure;
* Significant gastro-intestinal dysfunction;
* Varsity Athlete;
* Two or more previous concussions;
* Women who are pregnant or breast feeding;
* Taking tetracycline, fluoroquinolone, iron digoxin, chlorpromazine or penicillamine

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache Intensity and Duration | 14 days
  t-test of mean differences between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Hartman, MD, Principal Investigator — UVA Student Health and Wellness
Locations (1):
- University of Virginia Student Health and Wellness Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No